CLINICAL TRIAL: NCT01995292
Title: Comparative Clinical Trial of Conventional and Modified "Spray as You go" Technique With the "Enk Fiberoptic Atomizer Set" for Awake Fiberoptic Intubation (Atomizer Study)
Brief Title: Comparison of Two Different Types of "Spray as You go" Technique for Awake Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Nina Pirlich, Dr. med., Dr. med. Nina Pirlich, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Atomizer1.0
Record Dates: First submitted 2013-11-01; First posted 2013-11-26 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Awake Fiberoptic Intubation
Keywords: awake fiberoptic intubation; spray as you go technique; anesthesia; Enk Fiberoptic Atomizer Set
MeSH Terms: interventions — Bronchoscopes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- bronchoscope (Experimental): Patients will receive local anaesthetics via the working channel of the bronchoscope.
  Interventions: Device: bronchoscope
- Enk Fiberoptic Atomizer (Experimental): Patients will receive local anaesthetics for the awake fiberoptic intubation via the Enk Fiberoptic Atomizer.
  Interventions: Device: Enk Fiberoptic Atomizer

INTERVENTIONS:
Device: bronchoscope
  Other Names: Standard procedure: Instillation of local anesthetics via the working channel of the bronchoscope
  Arms: bronchoscope
Device: Enk Fiberoptic Atomizer
  Other Names: Nebulization of local anesthetics with the Enk Fiberoptic Atomizer during awake fiberoptic intubation
  Arms: Enk Fiberoptic Atomizer

SUMMARY:
The purpose of this study is to determine whether modified "spray as you go" technique using the Enk Fiberoptic Atomizer Set during awake fiberoptic intubation is more comfortable for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* no concurrent participation in another clinical trial
* German language in speaking and writing
* Capability of giving consent
* written informed consent
* an elective surgery under general anesthesia, in which an awake fiberoptic intubation is indicated

Exclusion Criteria:

* Age < 18 years
* pregnant women
* patients unwilling or unable to give informed consent
* ASA classification > 3
* Known allergy to local anesthetics
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Comfort evaluation by the patient | up to 4 weeks
  Comparison of conventional and modified "spray as you go" technique

SECONDARY OUTCOMES:
Comfort evaluation by the performing as well as assisting anesthetist | up to 4 weeks
  Comparison of conventional and modified "spray as you go" technique
Comfort evaluation by the present nurses | up to 4 weeks
  Comparison of conventional and modified "spray as you go" technique
Patient response (coughing, gagging, grimacing, defenses) | up to 4 weeks
  Comparison of conventional and modified "spray as you go" technique
Vital signs | up to 4 weeks
  Comparison of conventional and modified "spray as you go" technique

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg - Universität, Mainz, Rhineland-Palatinate, Germany